CLINICAL TRIAL: NCT06405958
Title: Analysis of Microbiome Changes and Prognostic Association After Solid Organ Transplantation
Brief Title: Gut Microbiome Analysis in Organ Transplant Recipient
Status: Not yet recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Professor, Asan Medical Center
Other Study IDs: S2024-0859-0001
Record Dates: First submitted 2024-05-05; First posted 2024-05-09 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Microbial Colonization
Keywords: microbiota; solid organ transplantation; metagenomic sequencing
MeSH Terms: conditions — Communicable Diseases | interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Enrollment of liver, kidney, heart, pancreas, and lung solid organ transplant recipients and regular collection of stool samples (at the time of transplantation, 1 month, 6~12months after transplantation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Liver transplant patients: Patients who have undergone liver transplantation
  Interventions: Other: gut microbiome
- Kidney transplant patients: Patients who have undergone kidney transplantation
  Interventions: Other: gut microbiome
- Pancreas transplant patients: Patients who have undergone pancreas transplantation
  Interventions: Other: gut microbiome
- Heart transplant patients: Patients who have undergone heart transplantation
  Interventions: Other: gut microbiome
- Lung transplant patients: Patients who have undergone lung transplantation
  Interventions: Other: gut microbiome

INTERVENTIONS:
Other: gut microbiome — Obtaining new gut microbiome data in organ transplantation

SUMMARY:
The microbiome acts as an antigen and can induce signaling through receptors like TLRs and NODs. Microbial metabolites can directly act on gut cells or reach other organs systemically. Studies show that the commensal, non-pathogenic microbiota plays an important role in regulating the immune system in various ways:

* Promoting differentiation of Th17 cells and ILC3 signaling to regulate IL-17A production
* Influencing iNKT cell generation early in life to prevent inflammatory activities
* Facilitating CD4+ T cell differentiation and balancing Th1/Th2 responses
* Inducing regulatory T cells (Tregs) that promote immune homeostasis
* Tregs in Peyer's patches help maintain a microbiome that supports homeostasis

The microbiome influences T cells, B cells and immune homeostasis. This has implications for transplantation, where modulating the microbiome could impact the graft's acceptance by affecting the recipient's immune cells that respond to the transplant.

In summary, it highlights the microbiome's role in immune regulation and the potential for leveraging this interaction therapeutically, including in the context of transplantation.

DETAILED DESCRIPTION:
The microorganisms coexisting in our bodies are known to be involved in immune functions in various ways. The microbiome basically acts as an antigen in the immune system and is known to be able to induce ligands for toll-like receptors (TLRs) and NOD, which is one of the pattern recognition receptors. Microbial metabolites such as short-chain fatty acids (SCFAs) or AhR ligands can directly act on intestinal cells and gut immune cells, but can also reach other organs through systemic circulation and regulate immunity. Many studies have shown that not pathogenic but coexisting microbiota can regulate the immune system, as described below.

Intestinal colonization of segmented filamentous bacteria promotes the differentiation of CD4+Th17 cells and induces signaling through the ILC3/IL-22/SAA1/2 axis, leading to IL-17A production by RORγt+Th17 cells. IL-22 derived from ILC3 facilitates IL-17A production by Th17 cells, contributing to the inhibition of certain microbial species. Decreased MHCII expression in ILC3 prevents the activation of commensal-specific CD4+ T cells, avoiding immune responses against the colonization of harmless microbes. Early-life microbial colonization partially inhibits the generation of abundant iNKT cells through sphingolipid production, preventing potential disease-promoting activities in the intestinal lamina propria and lungs.

Colonization by Bacteroides fragilis, a major constituent of the mammalian gut microbiota, promotes CD4+ T cell differentiation and contributes to balancing Th1 and Th2 in a polysaccharide A-dependent manner. Polysaccharide A is taken up by lamina propria dendritic cells via TLR2 and presented to naive CD4+ T cells, which differentiate into regulatory T cells (iTregs) in the presence of active TGF-β, and the IL-10 produced by these cells promotes immune homeostasis.

Maintaining this immune homeostasis also requires selectively maintaining appropriate gut microbes. Foxp3+ Tregs contributing to immune homeostasis are located in Peyer's patches and induce class switching in B cells, thereby maintaining and managing a microbial composition that can sustain bodily homeostasis.

The above results exemplify how the immune system and the coexisting microbial ecosystem influence each other. This suggests that after transplantation, the microbiome can affect T cells, B cells, and consequently impact and be impacted by the graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received or are receiving solid organ transplants (liver, kidney, pancreas, heart, lung) at this hospital.
* Patients who have listened to and understood a detailed explanation of this study, and have voluntarily decided to participate and provided written consent.

Exclusion Criteria:

* Patients undergoing re-transplantation.
* Patients with a history of previous organ transplantation, except for cases where a pancreas transplant is performed after a kidney transplant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For liver transplant patients, 90 samples are expected with stool, blood, and saliva collection at baseline, 1 month, and 6-12 months post-transplant. 16S full-length sequencing will be performed on these samples. For kidney transplant recipients, 70 stool samples will undergo the same collection timing and 16S analysis. Heart transplant patients will contribute 10 stool samples following the same timepoints for 16S sequencing and RNA sequencing. Lung transplant recipients will provide 15 stool and blood samples at those timepoints for 16S full-length and RNA sequencing analysis. Finally, 15 stool and blood samples will be collected from pancreas transplant recipients per the stated schedule for 16S analysis only. The comprehensive sampling strategy across different organ groups aims to characterize microbiome and transcriptomic changes over the transplant period using appropriate molecular profiling methods.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the gut Microbiome | 3 years
  Collecting admission and regular stool samples from solid organ transplant recipients (liver, kidney, heart, pancreas, lung) and performing high-resolution microbiome analysis (based on 16S full-length sequencing) to investigate changes in the gut microbiome following transplantation and develop models to predict outcomes in these patients.